CLINICAL TRIAL: NCT03887117
Title: A Randomized, Controlled, Open-label, 4-arm Parallel Group Study to Evaluate the Effect of Switching From Cigarette Smoking to the Use of IQOS in Healthy Adult Current Smokers on Exercise Capacity and Trainability
Brief Title: Effect of Switching From Cigarette Smoking to IQOS on Exercise Capacity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philip Morris Products S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: P1-EXC-01-EU
Record Dates: First submitted 2019-02-28; First posted 2019-03-22 (Actual); Results first posted 2021-12-27 (Actual); Last update posted 2021-12-27 (Actual); Status verified 2021-11

CONDITIONS: Smoking; Exercise Capacity
Keywords: IQOS; Heated Tobacco
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- IQOS-1 (Active Comparator): IQOS + Exercise Training Program
  Subjects randomized to IQOS use will switch to IQOS use and participate in an exercise training program.
  Interventions: Other: IQOS + Exercise Training Program
- IQOS-2 (Active Comparator): IQOS without Exercise Training Program
  Subjects randomized to IQOS use will switch to IQOS use, but will not participate in an exercise training program.
  Interventions: Other: IQOS without Exercise Training Program
- Cigarette Smoking (Active Comparator): Cigarette Smoking + Exercise Training Program
  Subjects randomized to continued cigarette smoking and participation in an exercise training program.
  Interventions: Other: Cigarette Smoking + Exercise Training Program
- Smoking Abstinence (Active Comparator): Smoking Abstinence + Exercise Training Program
  Subjects randomized to smoking abstinence and participation in an exercise training program.
  Interventions: Other: Smoking Abstinence + Exercise Training Program

INTERVENTIONS:
Other: IQOS + Exercise Training Program — Switch to IQOS use + participation in a training program
  Arms: IQOS-1
Other: IQOS without Exercise Training Program — Switch to IQOS use only, without participation in a training program
  Arms: IQOS-2
Other: Cigarette Smoking + Exercise Training Program — Continue to smoke cigarettes + participation in a training program
  Arms: Cigarette Smoking
Other: Smoking Abstinence + Exercise Training Program — Switch to smoking abstinence + participation in a training program
  Arms: Smoking Abstinence

SUMMARY:
This exploratory study is part of the global clinical assessment program of IQOS. It was designed to provide scientific evidence to further substantiate the reduced risk potential of using a heated tobacco product (the Tobacco Heating System [THS] marketed as IQOS) as compared to smoking cigarettes. The main goals of this exploratory study were to assess whether switching from cigarette smoking to using IQOS would influence 1) maximum oxygen uptake during incremental exercise (VO2max) and exercise capacity, 2) ability to perform exercise training and thereby influence 3) VO2max after 12 weeks of exercise training, 4) physiological parameters and biological health markers, and finally 5) physical activity levels in daily life.

DETAILED DESCRIPTION:
This exploratory study, with healthy adult smokers, was designed without product use restrictions (ad libitum product use) in order to replicate as closely as possible "real life" conditions. Subjects randomized to the cigarette and IQOS arms were asked to buy their own cigarettes or HeatSticks, respectively. Subjects randomized to the smoking abstinence (SA) arm were instructed to stay smoking abstinent until the end of the study. Subjects in the SA arm received smoking abstinence support and, in order to prevent relapse to cigarette smoking during the training program, were also allowed to use nicotine replacement therapy.

Mobile health technology was used in the study to explore the impact on switching from smoking to using IQOS on physical activity in daily real-world living conditions. The wearable enabled non-invasive recording of physical activity in an objective manner throughout the study. However, results collected from this device will be reported separately.

It should be noted that some study outcomes were reported graphically, rather than numerically. Consequently, these outcomes have not been included in this results disclosure.

ELIGIBILITY:
Inclusion Criteria:

* Smoking, healthy subject based on safety laboratory, ECG, spirometry, vital signs, physical examination, medical history and Investigator's assessment.
* Subject has been smoking for at least three years prior to V1.
* Subject has been smoking ≥ 10 cigarettes per day over the last 12 months. Smoking status will be verified by a urinary cotinine ≥ 200 ng/mL and CO exhaled breath test > 10 ppm both at V1 and V2.
* Subject does not plan to quit smoking within 6 months after V1.

Exclusion Criteria:

* Subject has a clinically relevant disease which requires medication (including but not limited to gastrointestinal, renal, hepatic, neurological, hematological, endocrine, oncological, urological, immunological, pulmonary [such as but not limited to pulmonary oedema, asthma], and cardiovascular [such as, but not limited to myocardial infarction, unstable angina, uncontrolled arrhythmias, heart failure], disease) or any other clinically significant medical condition (including abnormal safety laboratory result as per CTCAE), which as per the judgment of the Investigator would jeopardize the safety of the subject.
* Subject performs more than 45 min of vigorous physical activity per week.
* Subject takes medication influencing blood volume such as erythropoietin, diuretics and beta blockers, or diabetic medications.
* Subject cannot participate in the study for any reason other than medical as per the Investigator's judgment (e.g. psychological and/or social reason)
* For women only: subject is pregnant (does not have negative pregnancy tests at V1 and at V2) or is breastfeeding.
* For women of childbearing potential : female subject who does not agree to using an acceptable method of effective contraception during the entire study.
* Subject has a BMI < 18.5 kg/m2 or BMI ≥ 30 kg/m2.
* Subject has a positive urine drug screen.
* Subject has been previously screened for this study.
* Subject, or one of their family members (e.g., spouse, parent, sibling or child), is a current or former employee of the tobacco industry.
* Subject, or one of their family members (e.g. spouse, parent, sibling or child), is an employee of the investigational site or any other parties involved in the study.
* Subject is legally incompetent, or physically or mentally incapable of giving consent (e.g., emergency situation, under guardianship, prisoners, or subjects who are involuntarily incarcerated).

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-11-25 (Actual); Study Completion 2020-03-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Armin Schultz, MD, Principal Investigator — CRS Clinical Research Services Mannheim GmbH; Christelle Haziza, PhD, Study Chair — Philip Morris Products S.A.
Locations (1):
- CRS Clinical Research Services Mannheim GmbH, Mannheim, Germany

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 94 subjects were enrolled into the study, but 1 subject was not randomized. 26 subjects were randomized to Cigarette arm, 25 subjects were randomized to IQOS-1 arm, 15 subjects to IQOS-2 arm, and 27 subjects to the Smoking Abstinence (SA) arm.
  Subjects were requested to use the product allocated to their respective study arm, but it was considered acceptable that not all subjects randomized to the IQOS arms or to the cigarette arm exclusively used the randomized product during the study.
Groups:
- IQOS-1: IQOS + Exercise Training Program
  Subjects randomized to IQOS use will switch to IQOS use and participate in an exercise training program.
  IQOS + Exercise Training Program: Switch to IQOS use + participation in a training program
- Cigarette Smoking: Cigarette Smoking + Exercise Training Program
  Subjects randomized to continued cigarette smoking and participation in an exercise training program.
  Cigarette Smoking + Exercise Training Program: Continue to smoke cigarettes + participation in a training program
- Smoking Abstinence: Smoking Abstinence + Exercise Training Program
  Subjects randomized to smoking abstinence and participation in an exercise training program.
  Smoking Abstinence + Exercise Training Program: Switch to smoking abstinence + participation in a training program
Period: Overall Study
Arm/Group | IQOS-1 | IQOS-2 | Cigarette Smoking | Smoking Abstinence
Started | 25 | 15 | 26 | 27
Completed | 25 | 14 | 25 | 25
Not Completed | 0 | 1 | 1 | 2
Not completed — Discontinued prematurely | 0 | 1 | 1 | 2

BASELINE CHARACTERISTICS:
Population: Full Analysis Set
Groups:
- IQOS-2: No Training
  Subjects randomized to IQOS use will switch to IQOS use, but will not participate in an exercise training program.
  No Training: Switch to IQOS use only, without participation in a training program
- Total: Total of all reporting groups
Arm/Group | IQOS-1 | IQOS-2 | Cigarette Smoking | Smoking Abstinence | Total
Number analyzed (Participants) | 24 | 14 | 25 | 27 | 90
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.8 (12.8) | 40.5 (13.4) | 40.0 (10.9) | 40.2 (10.3) | 39.8 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 7 | 14 | 16 | 49
  Male | 12 | 7 | 11 | 11 | 41
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 24 | 14 | 25 | 27 | 90
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Height (cm) [Mean (Standard Deviation); unit: cm] | 171 (10.3) | 171 (10.4) | 171 (8.25) | 171 (9.19) | 171 (9.27)
Cigarettes smoked/day (last year) [Mean (Standard Deviation); unit: cigarettes/day] | 18.8 (5.51) | 17.2 (4.3) | 18.0 (4.69) | 18.9 (6.66) | 18.4 (5.46)

OUTCOME MEASURES:

1. Primary Outcome: Maximal Oxygen Uptake (VO2max, Absolute Values)
Description: To measure VO2max during maximal cycle ergometer exercise (expressed in absolute values [mL*min-1]).
Time Frame: Measured at baseline (V3), at week 1 (V4), and at week 12 (V43).
Population: AEECS: As Exposed Exercise Compliant Set. Some participants were excluded from analysis for protocol deviations (including, but not limited to, missing measurements).
Measure: Mean (95% Confidence Interval); unit: mL/min
Groups:
- Dual-1: Subject randomized to IQOS-1 using ≥30 HeatSticks /month and ≥30 cigarettes/month.
- Dual-2: Subject randomized to IQOS-2 using ≥30 HeatSticks /month and ≥30 cigarettes/month.
- Other: Other (use of <30 HeatSticks/month and 5-30 cig/month or other forms of product use)
Arm/Group | Cigarette Smoking | IQOS-1 | IQOS-2 | Smoking Abstinence | Dual-1 | Dual-2 | Other
Number analyzed (Participants) | 21 | 19 | 13 | 22 | 1 | 1 | 8
mL/min
  Acute Baseline (V3): number analyzed (Participants) | 20 | 17 | 13 | 20 | 1 | 1 | 8
  Acute Baseline (V3) | 1878 [1715 to 2040] | 2027 [1799 to 2255] | 2197 [1788 to 2605] | 1950 [1708 to 2191] | 2750 | 1620 | 2103 [1775 to 2430]
  Acute Effect (V4): number analyzed (Participants) | 20 | 17 | 13 | 20 | 1 | 1 | 8
  Acute Effect (V4) | 1823 [1686 to 1960] | 2062 [1823 to 2300] | 2156 [1747 to 2565] | 2071 [1791 to 2351] | 2770 | 1770 | 2094 [1721 to 2466]
  Training Effect (V43): number analyzed (Participants) | 21 | 19 | 12 | 21 | 0 | 0 | 5
  Training Effect (V43) | 1977 [1807 to 2147] | 2178 [1889 to 2468] | 2150 [1709 to 2591] | 2292 [1984 to 2601] |  |  | 2182 [1628 to 2736]

2. Primary Outcome: Maximal Oxygen Uptake (VO2max, Weight-adjusted Values)
Description: To measure VO2max during maximal cycle ergometer exercise (expressed in weight-adjusted [mL*kg-1*min-1] values).
Time Frame: Measured at baseline (V3), at week 1 (V4), and at week 12 (V43).
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: mL/(kg*min)
Arm/Group | Cigarette Smoking | IQOS-1 | IQOS-2 | Smoking Abstinence | Dual-1 | Dual-2 | Other
Number analyzed (Participants) | 21 | 19 | 13 | 22 | 1 | 1 | 8
mL/(kg*min)
  Acute Baseline (V3): number analyzed (Participants) | 20 | 17 | 13 | 20 | 1 | 1 | 8
  Acute Baseline (V3) | 27.3 [24.8 to 29.8] | 27.4 [24.9 to 29.9] | 28.9 [24.6 to 33.3] | 25.1 [22.9 to 27.3] | 34.7 | 24.4 | 25.8 [21.8 to 29.8]
  Acute Effect (V4): number analyzed (Participants) | 20 | 17 | 13 | 20 | 1 | 1 | 8
  Acute Effect (V4) | 26.6 [24.4 to 28.8] | 27.9 [25.1 to 30.7] | 28.2 [24.4 to 32.0] | 26.7 [24.0 to 29.4] | 34.5 | 27.0 | 25.4 [21.3 to 29.5]
  Training Effect (V43): number analyzed (Participants) | 21 | 19 | 12 | 21 | 0 | 0 | 5
  Training Effect (V43) | 27.9 [25.1 to 30.8] | 28.8 [25.7 to 31.8] | 27.7 [23.1 to 32.3] | 29.6 [26.4 to 32.7] |  |  | 30.9 [27.9 to 34.0]

3. Primary Outcome: Maximal Oxygen Uptake (VO2max, Fat-free Weight Adjusted Values)
Description: To measure VO2max during maximal cycle ergometer exercise (expressed in fat-free weight adjusted values [mL*kg-1*min-1]).
Time Frame: Measured at baseline (V3), at week 1 (V4), and at week 12 (V43).
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: mL/(kg*min)
Arm/Group | Cigarette Smoking | IQOS-1 | IQOS-2 | Smoking Abstinence | Dual-1 | Dual-2 | Other
Number analyzed (Participants) | 21 | 19 | 13 | 22 | 1 | 1 | 8
mL/(kg*min)
  Acute Baseline (V3): number analyzed (Participants) | 20 | 17 | 13 | 20 | 1 | 1 | 8
  Acute Baseline (V3) | 37.5 [34.4 to 40.5] | 38.4 [35.3 to 41.6] | 38.3 [34.0 to 42.6] | 34.8 [32.7 to 36.9] | 44.1 | 34.3 | 34.4 [29.5 to 39.3]
  Acute Effect (V4): number analyzed (Participants) | 20 | 17 | 13 | 20 | 1 | 1 | 8
  Acute Effect (V4) | 37.0 [33.8 to 40.2] | 39.8 [35.6 to 44.0] | 37.6 [34.3 to 41.0] | 37.0 [34.6 to 39.5] | 45.3 | 40.2 | 34.1 [30.1 to 38.1]
  Training Effect (V43): number analyzed (Participants) | 21 | 19 | 12 | 21 | 0 | 0 | 5
  Training Effect (V43) | 40.3 [36.4 to 44.2] | 39.8 [36.5 to 43.1] | 38.1 [34.4 to 41.8] | 42.0 [38.7 to 45.2] |  |  | 44.7 [36.2 to 53.1]

4. Primary Outcome: Exercise Capacity
Description: To measure exercise capacity, by measuring time to complete a pre-defined work (determined as 25% more work than the study subject produced during baseline VO2max test) on a cycle ergometer (seconds).
Time Frame: Measured at baseline (V3), at week 1 (V4), and at week 12 (V43)
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: seconds
Arm/Group | Cigarette Smoking | IQOS-1 | IQOS-2 | Smoking Abstinence | Dual-1 | Dual-2 | Other
Number analyzed (Participants) | 21 | 19 | 13 | 22 | 1 | 1 | 8
seconds
  Acute Baseline (V3): number analyzed (Participants) | 19 | 17 | 13 | 20 | 1 | 1 | 8
  Acute Baseline (V3) | 2283 [2033 to 2534] | 2366 [2109 to 2623] | 2330 [2013 to 2648] | 2156 [1975 to 2337] | 2110 | 2871 | 2147 [1722 to 2571]
  Acute Effect (V4): number analyzed (Participants) | 19 | 14 | 12 | 19 | 1 | 1 | 8
  Acute Effect (V4) | 2205 [2017 to 2394] | 2189 [1949 to 2429] | 2170 [1877 to 2462] | 2210 [1921 to 2498] | 2402 | 3006 | 2190 [1820 to 2561]
  Training Effect (V43): number analyzed (Participants) | 19 | 18 | 11 | 21 | 0 | 0 | 4
  Training Effect (V43) | 1985 [1728 to 2242] | 2123 [1926 to 2319] | 2374 [1970 to 2777] | 1849 [1623 to 2075] |  |  | 1982 [1465 to 2498]

5. Primary Outcome: Exercise Training Intensity: Cumulative Work
Description: To measure cumulative work (calories) produced during each 40 minute exercise training session, performed on a stationary bike, over 12 weeks.
Time Frame: Measured during 38 exercise training sessions of 40 minutes duration, conducted approximately 3 times a week, over 12 weeks.
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: calorie
Arm/Group | Cigarette Smoking | IQOS-1 | Smoking Abstinence | Other
Number analyzed (Participants) | 21 | 19 | 22 | 5
calorie
  Baseline (V5): number analyzed (Participants) | 21 | 19 | 21 | 4
  Baseline (V5) | 169 [145 to 193] | 222 [196 to 249] | 208 [176 to 239] | 203 [108 to 297]
  V14: number analyzed (Participants) | 21 | 18 | 22 | 4
  V14 | 203 [175 to 231] | 196 [167 to 226] | 231 [200 to 261] | 195 [135 to 255]
  V29: number analyzed (Participants) | 21 | 19 | 22 | 3
  V29 | 183 [155 to 211] | 197 [159 to 235] | 223 [196 to 249] | 214 [186 to 243]
  V41: number analyzed (Participants) | 20 | 18 | 20 | 3
  V41 | 187 [161 to 212] | 199 [169 to 230] | 211 [183 to 239] | 219 [80.5 to 357]

6. Primary Outcome: Exercise Training Intensity: Average Work Rate
Description: To measure the average work rate (watt) during each 40 minute exercise training session, performed on a stationary bike, over 12 weeks.
Time Frame: as for outcome 5
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Watt
Arm/Group | Cigarette Smoking | IQOS-1 | Smoking Abstinence | Other
Number analyzed (Participants) | 21 | 19 | 22 | 5
Watt
  Baseline (V5): number analyzed (Participants) | 21 | 19 | 21 | 4
  Baseline (V5) | 70.7 [61.1 to 80.3] | 87.6 [77.2 to 98.0] | 84.4 [71.1 to 97.8] | 82.8 [44.9 to 121]
  V14: number analyzed (Participants) | 21 | 18 | 22 | 4
  V14 | 81.7 [69.8 to 93.7] | 78.7 [66.9 to 90.6] | 90.5 [78.3 to 103] | 80.5 [55.4 to 106]
  V29: number analyzed (Participants) | 21 | 19 | 22 | 3
  V29 | 74.0 [63.1 to 84.8] | 80.4 [64.7 to 96.2] | 90.9 [80.3 to 101] | 85.3 [54.5 to 116]
  V41: number analyzed (Participants) | 20 | 18 | 20 | 3
  V41 | 76.9 [66.3 to 87.5] | 82.1 [69.4 to 94.8] | 85.8 [74.0 to 97.5] | 89.0 [29.2 to 149]

7. Primary Outcome: Exercise Training Intensity: Average Heart Rate
Description: To measure the average heart rate (bpm) during each 40 minute exercise training session, performed on a stationary bike, over 12 weeks.
Time Frame: as for outcome 5
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: beats/minute
Arm/Group | Cigarette Smoking | IQOS-1 | Smoking Abstinence | Other
Number analyzed (Participants) | 21 | 19 | 22 | 5
beats/minute
  Baseline (V5): number analyzed (Participants) | 21 | 19 | 21 | 4
  Baseline (V5) | 125 [119 to 131] | 127 [122 to 132] | 123 [117 to 128] | 110 [77.7 to 142]
  V14: number analyzed (Participants) | 21 | 18 | 22 | 4
  V14 | 119 [108 to 130] | 127 [121 to 133] | 121 [117 to 126] | 125 [120 to 130]
  V29: number analyzed (Participants) | 21 | 19 | 22 | 3
  V29 | 124 [116 to 131] | 124 [118 to 130] | 121 [116 to 125] | 123 [113 to 133]
  V41: number analyzed (Participants) | 20 | 18 | 20 | 3
  V41 | 125 [119 to 130] | 122 [115 to 130] | 123 [118 to 128] | 120 [98.0 to 141]

8. Primary Outcome: Exercise Training Intensity: Time Spent at Maximal Heart Rate
Description: To measure the time (seconds) spent at 0-50%, 50-60%, 60-70%, 70-80 % and >80% of maximal heart rate during each 40 minute exercise training session, performed on a stationary bike, over 12 weeks.
Time Frame: as for outcome 5
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: seconds
Arm/Group | Cigarette Smoking | IQOS-1 | Smoking Abstinence | Other
Number analyzed (Participants) | 21 | 19 | 22 | 5
seconds
  V5 (Baseline): 0-50%: number analyzed (Participants) | 19 | 19 | 21 | 4
  V5 (Baseline): 0-50% | 33.7 [1.00 to 66.4] | 26.1 [-7.68 to 59.8] | 14.2 [-2.15 to 30.5] | 361 [-346 to 1068]
  V5 (Baseline): 50-60%: number analyzed (Participants) | 19 | 19 | 21 | 4
  V5 (Baseline): 50-60% | 29.7 [6.05 to 53.3] | 42.2 [14.7 to 69.7] | 38.6 [18.3 to 58.9] | 162 [-154 to 479]
  V5 (Baseline): 60-70%: number analyzed (Participants) | 19 | 19 | 21 | 4
  V5 (Baseline): 60-70% | 86.1 [43.8 to 128] | 130 [84.2 to 176] | 131 [78.0 to 184] | 301 [-242 to 843]
  V5 (Baseline): 70-80%: number analyzed (Participants) | 19 | 19 | 21 | 4
  V5 (Baseline): 70-80% | 793 [615 to 971] | 737 [586 to 888] | 743 [564 to 923] | 591 [378 to 803]
  V5 (Baseline): >80%: number analyzed (Participants) | 19 | 19 | 21 | 4
  V5 (Baseline): >80% | 1438 [1193 to 1683] | 1405 [1218 to 1591] | 1415 [1179 to 1650] | 944 [-372 to 2260]
  Visit 14: 0-50%: number analyzed (Participants) | 19 | 17 | 21 | 4
  Visit 14: 0-50% | 12.4 [0.479 to 24.4] | 7.24 [2.73 to 11.7] | 13.5 [4.26 to 22.8] | 7.0 [-15.3 to 29.3]
  Visit 14: 50-60%: number analyzed (Participants) | 19 | 17 | 21 | 4
  Visit 14: 50-60% | 25.3 [9.05 to 41.6] | 32.1 [15.0 to 49.3] | 38.0 [21.9 to 54.1] | 28.5 [-2.07 to 59.1]
  Visit 14: 60-70%: number analyzed (Participants) | 19 | 17 | 21 | 4
  Visit 14: 60-70% | 145 [22.7 to 267] | 139 [82.5 to 195] | 188 [80.8 to 295] | 77.8 [-50.1 to 206]
  Visit 14: 70-80%: number analyzed (Participants) | 19 | 17 | 21 | 4
  Visit 14: 70-80% | 807 [616 to 997] | 783 [606 to 960] | 880 [691 to 1068] | 888 [430 to 1346]
  Visit 14: >80%: number analyzed (Participants) | 19 | 17 | 21 | 4
  Visit 14: >80% | 1370 [1100 to 1641] | 1424 [1197 to 1650] | 1260 [993 to 1527] | 1386 [764 to 2007]
  Visit 29: 0-50%: number analyzed (Participants) | 20 | 19 | 22 | 3
  Visit 29: 0-50% | 83.1 [-62.7 to 229] | 17.2 [-0.0182 to 34.4] | 32.2 [-2.92 to 67.3] | 30.0 [-99.1 to 159]
  Visit 29: 50-60%: number analyzed (Participants) | 20 | 19 | 22 | 3
  Visit 29: 50-60% | 25.3 [-7.86 to 58.5] | 32.9 [4.18 to 61.7] | 43.0 [13.9 to 72.1] | 54.7 [-157 to 267]
  Visit 29: 60-70%: number analyzed (Participants) | 20 | 19 | 22 | 3
  Visit 29: 60-70% | 120 [42.8 to 197] | 236 [96.3 to 375] | 259 [65.8 to 453] | 130 [-277 to 538]
  Visit 29: 70-80%: number analyzed (Participants) | 20 | 19 | 22 | 3
  Visit 29: 70-80% | 731 [524 to 938] | 887 [690 to 1084] | 732 [544 to 920] | 855 [107 to 1604]
  Visit 29: >80%: number analyzed (Participants) | 20 | 19 | 22 | 3
  Visit 29: >80% | 1411 [1119 to 1704] | 1201 [933 to 1468] | 1293 [1032 to 1554] | 1286 [212 to 2360]
  Visit 41: 0-50%: number analyzed (Participants) | 18 | 17 | 20 | 3
  Visit 41: 0-50% | 11.1 [2.12 to 20.0] | 22.6 [-4.70 to 50.0] | 6.60 [1.12 to 12.1] | 1.33 [-4.40 to 7.07]
  Visit 41: 50-60%: number analyzed (Participants) | 18 | 17 | 20 | 3
  Visit 41: 50-60% | 12.3 [4.77 to 19.9] | 34.0 [3.49 to 64.5] | 25.5 [11.2 to 39.8] | 5.33 [-17.6 to 28.3]
  Visit 41: 60-70%: number analyzed (Participants) | 18 | 17 | 20 | 3
  Visit 41: 60-70% | 99.3 [51.0 to 148] | 308 [59.1 to 557] | 171 [84.6 to 257] | 271 [-685 to 1226]
  Visit 41: 70-80%: number analyzed (Participants) | 18 | 17 | 20 | 3
  Visit 41: 70-80% | 871 [609 to 1133] | 825 [607 to 1043] | 877 [621 to 1133] | 1032 [-86.6 to 2151]
  Visit 41: >80%: number analyzed (Participants) | 18 | 17 | 20 | 3
  Visit 41: >80% | 1377 [1066 to 1689] | 1185 [842 to 1528] | 1293 [968 to 1617] | 1091 [-999 to 3181]

9. Primary Outcome: Hemoglobin Mass
Description: To measure Hemoglobin mass (g), measured with the carbon monoxide-rebreathing method.
Time Frame: Measured at Baseline (V3) and week 12 (V43).
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: g
Arm/Group | Cigarette Smoking | IQOS-1 | IQOS-2 | Smoking Abstinence | Other
Number analyzed (Participants) | 21 | 19 | 13 | 22 | 5
g
  Baseline (V3): number analyzed (Participants) | 21 | 19 | 13 | 21 | 4
  Baseline (V3) | 861 [747 to 975] | 796 [701 to 891] | 905 [808 to 1003] | 883 [755 to 1012] | 766 [290 to 1241]
  Week 12 (V43): number analyzed (Participants) | 21 | 19 | 12 | 21 | 5
  Week 12 (V43) | 1194 [1001 to 1387] | 1176 [1005 to 1347] | 1224 [957 to 1490] | 1217 [966 to 1468] | 900 [454 to 1345]

10. Primary Outcome: Red Blood Cell Volume
Description: To measure Red blood cell volume (mL), measured with the carbon monoxide-rebreathing method.
Time Frame: Measured at Baseline (V3) and week 12 (V43).
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: mL
Arm/Group | Cigarette Smoking | IQOS-1 | IQOS-2 | Smoking Abstinence | Other
Number analyzed (Participants) | 21 | 19 | 13 | 22 | 5
mL
  Baseline (V3): number analyzed (Participants) | 21 | 19 | 13 | 21 | 4
  Baseline (V3) | 2541 [2207 to 2875] | 2353 [2076 to 2629] | 2681 [2388 to 2975] | 2605 [2231 to 2979] | 2269 [871 to 3667]
  Week 12 (V43): number analyzed (Participants) | 21 | 19 | 12 | 21 | 5
  Week 12 (V43) | 3523 [2959 to 4086] | 3478 [2988 to 3967] | 3618 [2838 to 4398] | 3605 [2900 to 4309] | 2623 [1357 to 3890]

11. Primary Outcome: Plasma Volume
Description: To measure Plasma volume (mL), measured with the carbon monoxide-rebreathing method.
Time Frame: Measured at Baseline (V3) and week 12 (V43).
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: mL
Arm/Group | Cigarette Smoking | IQOS-1 | IQOS-2 | Smoking Abstinence | Other
Number analyzed (Participants) | 21 | 19 | 13 | 22 | 5
mL
  Baseline (V3): number analyzed (Participants) | 21 | 19 | 13 | 21 | 4
  Baseline (V3) | 3429 [3044 to 3814] | 3156 [2811 to 3500] | 3558 [3242 to 3874] | 3521 [3075 to 3966] | 3252 [1558 to 4946]
  Week 12 (V43): number analyzed (Participants) | 21 | 19 | 12 | 21 | 5
  Week 12 (V43) | 4840 [4139 to 5542] | 4938 [4306 to 5570] | 4959 [4190 to 5729] | 5281 [4317 to 6245] | 4272 [2238 to 6307]

12. Primary Outcome: Total Blood Volume
Description: To measure total blood volume (mL), measured with the carbon monoxide-rebreathing method.
Time Frame: Measured at Baseline (V3) and week 12 (V43).
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: mL
Arm/Group | Cigarette Smoking | IQOS-1 | IQOS-2 | Smoking Abstinence | Other
Number analyzed (Participants) | 21 | 19 | 13 | 22 | 5
mL
  Baseline (V3): number analyzed (Participants) | 21 | 19 | 13 | 21 | 4
  Baseline (V3) | 5970 [5282 to 6657] | 5508 [4914 to 6102] | 6239 [5709 to 6770] | 6126 [5326 to 6925] | 5521 [2443 to 8599]
  Week 12 (V43): number analyzed (Participants) | 21 | 19 | 12 | 21 | 5
  Week 12 (V43) | 8363 [7151 to 9575] | 8416 [7334 to 9498] | 8577 [7060 to 10095] | 8886 [7263 to 10508] | 6896 [3618 to 10173]

13. Primary Outcome: Capillary Blood Lactate Levels
Description: To measure changes from baseline of Capillary blood lactate levels (mmol/L), measured (with a portable lactate analyzer) during VO2max test.
Time Frame: Measured at Baseline and week 15.
Reporting Status: Not Posted

14. Primary Outcome: Ventilation at VO2 Max
Description: To measure ventilation (L/min) at VO2max.
Time Frame: Measured at Baseline (V3), at week 1 (V4), and at week 12 (V43).
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: L/min
Arm/Group | Cigarette Smoking | IQOS-1 | IQOS-2 | Smoking Abstinence | Dual-1 | Dual-2 | Other
Number analyzed (Participants) | 21 | 19 | 13 | 22 | 1 | 1 | 8
L/min
  Baseline (V3): number analyzed (Participants) | 20 | 17 | 13 | 20 | 1 | 1 | 8
  Baseline (V3) | 74.8 [66.1 to 83.4] | 78.9 [70.4 to 87.4] | 87.3 [74.1 to 101] | 71.9 [65.9 to 77.8] | 109 | 55.7 | 77.2 [64.8 to 89.6]
  Acute Effect (V4): number analyzed (Participants) | 20 | 17 | 13 | 20 | 1 | 1 | 8
  Acute Effect (V4) | 72.0 [66.1 to 77.9] | 79.1 [70.4 to 87.9] | 81.3 [67.4 to 95.1] | 77.2 [69.0 to 85.5] | 110 | 78.6 | 76.1 [63.2 to 89.0]
  Training Effect (V43): number analyzed (Participants) | 21 | 19 | 12 | 21 | 0 | 0 | 5
  Training Effect (V43) | 72.7 [64.8 to 80.6] | 79.2 [69.8 to 88.6] | 82.5 [67.7 to 97.4] | 80.3 [73.6 to 87.1] |  |  | 72.0 [53.8 to 90.3]

15. Primary Outcome: Respiratory Rate
Description: To measure respiratory rate (breaths per minute) at VO2max.
Time Frame: Measured at Baseline (V3), at week 1 (V4), and at week 12 (V43).
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: breaths/minute
Arm/Group | Cigarette Smoking | IQOS-1 | IQOS-2 | Smoking Abstinence | Dual-1 | Dual-2 | Other
Number analyzed (Participants) | 21 | 19 | 13 | 22 | 1 | 1 | 8
breaths/minute
  Acute Baseline (V3): number analyzed (Participants) | 20 | 17 | 13 | 20 | 1 | 1 | 8
  Acute Baseline (V3) | 34.5 [31.3 to 37.7] | 37.5 [33.4 to 41.5] | 37.1 [30.7 to 43.4] | 35.2 [32.1 to 38.2] | 36.0 | 29.0 | 35.6 [32.3 to 39.0]
  Acute Effect (V4): number analyzed (Participants) | 20 | 17 | 13 | 20 | 1 | 1 | 8
  Acute Effect (V4) | 34.1 [30.4 to 37.7] | 37.8 [33.4 to 42.3] | 35.4 [32.0 to 38.8] | 36.1 [32.8 to 39.3] | 38.0 | 37.0 | 34.1 [30.0 to 38.2]
  Training Effect (V43: number analyzed (Participants) | 21 | 19 | 12 | 21 | 0 | 0 | 5
  Training Effect (V43 | 33.8 [30.4 to 37.2] | 37.0 [32.9 to 41.1] | 33.8 [30.4 to 37.3] | 36.3 [33.2 to 39.4] |  |  | 38.4 [29.7 to 47.1]

16. Primary Outcome: VCO2
Description: To measure VCO2 (L/min) at VO2 max.
Time Frame: Measured at Baseline (V3), at week 1 (V4), and at week 12 (V43).
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: L/min
Arm/Group | Cigarette Smoking | IQOS-1 | IQOS-2 | Smoking Abstinence | Dual-1 | Dual-2 | Other
Number analyzed (Participants) | 21 | 19 | 13 | 22 | 1 | 1 | 8
L/min
  Acute Baseline (V3): number analyzed (Participants) | 20 | 17 | 13 | 20 | 1 | 1 | 8
  Acute Baseline (V3) | 2.21 [2.01 to 2.42] | 2.36 [2.07 to 2.65] | 2.58 [2.14 to 3.02] | 2.24 [2.00 to 2.49] | 3.23 | 1.70 | 2.39 [1.98 to 2.80]
  Acute Effect (V4): number analyzed (Participants) | 20 | 17 | 13 | 20 | 1 | 1 | 8
  Acute Effect (V4) | 2.19 [2.01 to 2.36] | 2.41 [2.13 to 2.70] | 2.53 [2.04 to 3.02] | 2.41 [2.08 to 2.73] | 3.28 | 2.10 | 2.38 [1.98 to 2.78]
  Training Effect (V43): number analyzed (Participants) | 21 | 19 | 12 | 21 | 0 | 0 | 5
  Training Effect (V43) | 2.36 [2.12 to 2.59] | 2.53 [2.16 to 2.90] | 2.53 [2.01 to 3.05] | 2.67 [2.35 to 2.99] |  |  | 2.63 [1.96 to 3.29]

17. Primary Outcome: Respiratory Exchange Ratio
Description: To measure the respiratory exchange ratio (VCO2/VO2) at VO2max
Time Frame: Measured at Baseline (V3), at week 1 (V4), and at week 12 (V43).
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: ratio
Arm/Group | Cigarette Smoking | IQOS-1 | IQOS-2 | Smoking Abstinence | Dual-1 | Dual-2 | Other
Number analyzed (Participants) | 21 | 19 | 13 | 22 | 1 | 1 | 8
ratio
  Acute baseline (V3): number analyzed (Participants) | 20 | 17 | 13 | 20 | 1 | 1 | 8
  Acute baseline (V3) | 1.18 [1.14 to 1.22] | 1.16 [1.12 to 1.20] | 1.19 [1.14 to 1.23] | 1.16 [1.12 to 1.20] | 1.17 | 1.05 | 1.14 [1.05 to 1.23]
  Acute effect (V4): number analyzed (Participants) | 20 | 17 | 13 | 20 | 1 | 1 | 8
  Acute effect (V4) | 1.20 [1.15 to 1.25] | 1.17 [1.13 to 1.22] | 1.18 [1.15 to 1.21] | 1.17 [1.12 to 1.21] | 1.18 | 1.19 | 1.14 [1.06 to 1.21]
  Training Effect (V43): number analyzed (Participants) | 21 | 19 | 12 | 21 | 0 | 0 | 5
  Training Effect (V43) | 1.16 [1.11 to 1.21] | 1.16 [1.12 to 1.20] | 1.18 [1.14 to 1.22] | 1.18 [1.14 to 1.22] |  |  | 1.21 [1.14 to 1.27]

18. Primary Outcome: Rating of Perceived Capacity by Sex
Description: To measure Rating of Perceived Capacity (RPC), determined by using the RPC scale. The RPC scale is a list of physical activities arranged in order, with a scale of values from least strenuous (1) to most exhausting (18 for women, 20 for men). Subjects choose the most strenuous activity, with corresponding value, which they could sustain for 30 minutes.
Time Frame: Measured at Baseline (V3), at week 1 (V4), and at week 12 (V43).
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Rating of Perceived Capacity
Arm/Group | Cigarette Smoking | IQOS-1 | IQOS-2 | Smoking Abstinence | Dual-1 | Dual-2 | Other
Number analyzed (Participants) | 21 | 19 | 13 | 22 | 1 | 1 | 8
Rating of Perceived Capacity
  Acute Baseline - Female (V3): number analyzed (Participants) | 13 | 9 | 6 | 10 | 0 | 1 | 4
  Acute Baseline - Female (V3) | 7.77 [5.75 to 9.79] | 8.22 [6.56 to 9.89] | 8.17 [5.83 to 10.5] | 8.00 [7.11 to 8.89] |  | 5.00 | 8.50 [4.50 to 12.5]
  Acute Effect - Female (V4): number analyzed (Participants) | 13 | 9 | 6 | 10 | 0 | 1 | 4
  Acute Effect - Female (V4) | 7.15 [6.46 to 7.84] | 7.22 [5.31 to 9.14] | 7.83 [7.40 to 8.26] | 7.90 [6.34 to 9.46] |  | 5.00 | 8.50 [4.50 to 12.5]
  Acute Baseline - Male (V3): number analyzed (Participants) | 7 | 8 | 7 | 10 | 1 | 0 | 4
  Acute Baseline - Male (V3) | 8.00 [6.49 to 9.51] | 8.25 [7.28 to 9.22] | 9.71 [7.06 to 12.4] | 9.70 [7.85 to 11.5] | 8.00 |  | 7.00 [4.09 to 9.91]
  Acute Effect - Male (V4): number analyzed (Participants) | 7 | 8 | 7 | 10 | 1 | 0 | 4
  Acute Effect - Male (V4) | 6.86 [5.73 to 7.98] | 9.13 [7.68 to 10.6] | 10.7 [8.53 to 12.9] | 9.90 [8.53 to 11.3] | 9.00 |  | 6.25 [3.86 to 8.64]
  Training Baseline - Female (V3): number analyzed (Participants) | 12 | 9 | 6 | 11 | 0 | 0 | 5
  Training Baseline - Female (V3) | 6.92 [6.04 to 7.79] | 8.22 [6.56 to 9.89] | 7.67 [4.96 to 10.4] | 8.00 [7.21 to 8.79] |  |  | 10.4 [4.47 to 16.3]
  Training Effect - Female (V43): number analyzed (Participants) | 12 | 9 | 5 | 11 | 0 | 0 | 5
  Training Effect - Female (V43) | 8.58 [7.27 to 9.90] | 9.11 [7.55 to 10.7] | 8.60 [6.18 to 11.0] | 8.91 [7.49 to 10.3] |  |  | 9.60 [5.81 to 13.4]
  Training Baseline - Male (V3): number analyzed (Participants) | 9 | 10 | 7 | 11 | 0 | 0 | 0
  Training Baseline - Male (V3) | 7.67 [6.34 to 9.00] | 8.30 [7.54 to 9.06] | 9.71 [7.06 to 12.4] | 9.36 [7.55 to 11.2] |  |  |
  Training Effect - Male (V43): number analyzed (Participants) | 9 | 10 | 7 | 10 | 0 | 0 | 0
  Training Effect - Male (V43) | 8.33 [6.26 to 10.4] | 10.1 [8.69 to 11.5] | 9.14 [7.34 to 10.9] | 11.8 [9.24 to 14.4] |  |  |

19. Primary Outcome: Rating of Perceived Exertion
Description: To measure changes from baseline of the Rating of Perceived Exertion, determined by using the Borg scale. The Borg RPE scale is a numerical scale that ranges from 6 to 20, where 6 means "no exertion at all" and 20 means "maximal exertion." Subjects choose a number from the scale that best describes their level of exertion during a physical activity.
Time Frame: Measured at Baseline (V3), at week 1 (V4), and at week 12 (V43).
Reporting Status: Not Posted

20. Primary Outcome: Heart Rate
Description: To measure changes from baseline of heart rate (bpm) during VO2max test.
Time Frame: Measured at Baseline, at week 1, and at week 15.
Reporting Status: Not Posted

21. Primary Outcome: Oxygen Uptake
Description: To measure changes from baseline of Oxygen uptake during VO2max test. (mL/min)
Time Frame: Measured at Baseline, at week 1, and at week 15.
Reporting Status: Not Posted

22. Primary Outcome: High Density Lipoprotein (HDL)
Description: To measure HDL concentrations in serum (mg/dL).
Time Frame: Measured at Baseline (V3), week 6 (V14), week 10 (V28), and week 12 (V43).
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Cigarette Smoking | IQOS-1 | IQOS-2 | Smoking Abstinence | Other
Number analyzed (Participants) | 21 | 19 | 13 | 22 | 5
mg/dL
  Baseline (V3) | 49.3 [44.9 to 53.7] | 48.2 [40.3 to 56.0] | 47.1 [39.7 to 54.6] | 52.1 [45.6 to 58.7] | 55.4 [48.0 to 62.7]
  Week 6 (V14) | 48.6 [43.8 to 53.4] | 53.3 [45.5 to 61.1] | 51.0 [41.5 to 60.4] | 53.6 [47.4 to 59.7] | 54.7 [47.5 to 61.9]
  Week 10 (V28) | 51.0 [47.5 to 54.4] | 49.0 [41.1 to 57.0] | 51.8 [43.6 to 60.1] | 53.3 [45.9 to 60.7] | 56.2 [47.2 to 65.2]
  Week 12 (V43): number analyzed (Participants) | 21 | 19 | 12 | 21 | 5
  Week 12 (V43) | 47.8 [43.2 to 52.4] | 48.7 [41.2 to 56.2] | 50.1 [40.8 to 59.5] | 55.6 [49.6 to 61.7] | 49.1 [44.0 to 54.2]

23. Primary Outcome: Low Density Lipoprotein (LDL)
Description: To measure LDL concentrations in serum (mg/dL).
Time Frame: Measured at Baseline (V3), week 6 (V14), week 10 (V28), and week 12 (V43).
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Cigarette Smoking | IQOS-1 | IQOS-2 | Smoking Abstinence | Other
Number analyzed (Participants) | 21 | 19 | 13 | 22 | 5
mg/dL
  Baseline (V3) | 124 [107 to 141] | 111 [102 to 121] | 122 [109 to 136] | 115 [97.9 to 133] | 155 [101 to 208]
  Week 6 (V14) | 127 [112 to 142] | 108 [98.8 to 118] | 126 [106 to 145] | 104 [87.3 to 121] | 136 [79.4 to 193]
  Week 10 (V28) | 131 [115 to 148] | 105 [94.4 to 116] | 122 [105 to 138] | 106 [90.0 to 122] | 140 [104 to 176]
  Week 12 (V43): number analyzed (Participants) | 21 | 19 | 12 | 21 | 5
  Week 12 (V43) | 133 [111 to 155] | 105 [91.6 to 118] | 118 [101 to 135] | 109 [90.5 to 127] | 123 [81.5 to 164]

24. Primary Outcome: Very Low Density Lipoprotein (VLDL)
Description: To measure VLDL concentrations in serum (mg/dL).
Time Frame: Measured at Baseline (V3), week 6 (V14), week 10 (V28), and week 12 (V43).
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Cigarette Smoking | IQOS-1 | IQOS-2 | Smoking Abstinence | Other
Number analyzed (Participants) | 21 | 19 | 13 | 22 | 5
mg/dL
  Baseline (V3) | 14.7 [9.05 to 20.4] | 13.7 [8.29 to 19.1] | 15.8 [10.2 to 21.4] | 13.7 [8.45 to 18.9] | 12.5 [-1.89 to 26.9]
  Week 6 (V14) | 15.6 [5.38 to 25.8] | 8.30 [5.42 to 11.2] | 11.1 [5.63 to 16.6] | 11.4 [6.64 to 16.1] | 9.82 [4.76 to 14.9]
  Week 10 (V28): number analyzed (Participants) | 20 | 18 | 11 | 21 | 5
  Week 10 (V28) | 14.7 [9.06 to 20.4] | 13.7 [0.242 to 27.1] | 12.0 [6.79 to 17.1] | 6.56 [4.86 to 8.25] | 10.3 [5.21 to 15.4]
  Week 12 (V43): number analyzed (Participants) | 18 | 17 | 12 | 18 | 5
  Week 12 (V43) | 10.7 [7.41 to 13.9] | 12.4 [5.34 to 19.5] | 12.1 [6.31 to 18.0] | 12.3 [4.87 to 19.8] | 10.8 [5.91 to 15.6]

25. Primary Outcome: High Sensitivity C-reactive Protein (Hs-CRP)
Description: To measure hs-CRP concentrations in serum (mg/dL).
Time Frame: Measured at Baseline (V3), week 6 (V14), week 10 (V28), and week 12 (V43).
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: mg/L
Arm/Group | Cigarette Smoking | IQOS-1 | IQOS-2 | Smoking Abstinence | Other
Number analyzed (Participants) | 21 | 19 | 13 | 22 | 5
mg/L
  Baseline (V3) | 2.10 [0.590 to 3.62] | 2.19 [0.983 to 3.40] | 0.804 [0.432 to 1.18] | 1.80 [0.964 to 2.63] | 1.17 [-0.754 to 3.09]
  Week 6 (V14) | 1.40 [0.805 to 2.00] | 1.84 [0.845 to 2.83] | 1.24 [0.644 to 1.83] | 1.43 [0.833 to 2.03] | 1.37 [-0.729 to 3.47]
  Week 10 (V28) | 1.67 [1.11 to 2.23] | 2.57 [1.06 to 4.07] | 0.815 [0.438 to 1.19] | 2.38 [0.659 to 4.10] | 1.43 [-0.947 to 3.81]
  Week 12 (V43): number analyzed (Participants) | 21 | 19 | 12 | 21 | 5
  Week 12 (V43) | 1.55 [0.624 to 2.47] | 2.79 [0.399 to 5.19] | 1.69 [0.205 to 3.17] | 1.61 [0.745 to 2.48] | 1.26 [-1.08 to 3.60]

26. Primary Outcome: Growth Hormone
Description: To measure growth hormone concentrations in serum (ng/mL).
Time Frame: Measured at Baseline (V3), week 6 (V14), week 10 (V28), and week 12 (V43).
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Cigarette Smoking | IQOS-1 | IQOS-2 | Smoking Abstinence | Other
Number analyzed (Participants) | 21 | 19 | 13 | 22 | 5
ng/mL
  Baseline (V3) | 2.15 [0.726 to 3.58] | 1.37 [0.594 to 2.15] | 2.49 [0.0590 to 4.93] | 4.03 [0.381 to 7.67] | 2.02 [-1.36 to 5.41]
  Week 6 (V14) | 1.25 [0.452 to 2.06] | 1.49 [0.535 to 2.44] | 1.22 [0.333 to 2.10] | 1.30 [0.444 to 2.16] | 1.13 [-1.24 to 3.50]
  Week 10 (V28) | 1.45 [0.689 to 2.22] | 0.907 [0.394 to 1.42] | 1.31 [0.453 to 2.17] | 1.97 [0.729 to 3.21] | 0.536 [0.0523 to 1.02]
  Week 12 (V43): number analyzed (Participants) | 21 | 19 | 12 | 21 | 5
  Week 12 (V43) | 1.98 [0.487 to 3.47] | 1.44 [0.391 to 2.50] | 1.94 [0.175 to 3.70] | 1.55 [0.582 to 2.51] | 0.492 [0.0520 to 0.932]

27. Primary Outcome: Hemoglobin A1c (HbA1c)
Description: To measure glycosylated hemoglobin (HbA1c in whole blood).
Time Frame: Measured at Baseline (V3), week 6 (V14), week 10 (V28), and week 12 (V43).
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: % (of red blood cells)
Arm/Group | Cigarette Smoking | IQOS-1 | IQOS-2 | Smoking Abstinence | Other
Number analyzed (Participants) | 21 | 19 | 13 | 22 | 5
% (of red blood cells)
  Baseline (V3) | 5.44 [5.34 to 5.53] | 5.39 [5.27 to 5.51] | 5.38 [5.22 to 5.53] | 5.53 [5.37 to 5.68] | 5.36 [4.91 to 5.81]
  Week 6 (V14) | 5.41 [5.30 to 5.52] | 5.35 [5.21 to 5.49] | 5.41 [5.23 to 5.58] | 5.50 [5.34 to 5.66] | 5.28 [4.90 to 5.66]
  Week 10 (V28) | 5.38 [5.27 to 5.49] | 5.34 [5.22 to 5.46] | 5.38 [5.18 to 5.57] | 5.49 [5.32 to 5.65] | 5.28 [5.00 to 5.56]
  Week 12 (V43): number analyzed (Participants) | 21 | 19 | 12 | 21 | 5
  Week 12 (V43) | 5.40 [5.30 to 5.49] | 5.35 [5.22 to 5.47] | 5.34 [5.17 to 5.51] | 5.50 [5.34 to 5.66] | 5.34 [4.94 to 5.74]

28. Primary Outcome: Resting Systolic Blood Pressure
Description: To measure resting systolic blood pressure in mmHg.
Time Frame: Measured at Baseline (V3), week 6 (V14), week 10 (V28), and week 12 (V43).
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Cigarette Smoking | IQOS-1 | IQOS-2 | Smoking Abstinence | Other
Number analyzed (Participants) | 21 | 19 | 13 | 22 | 5
mmHg
  Baseline (V3) | 118 [113 to 123] | 121 [116 to 127] | 118 [110 to 126] | 122 [116 to 129] | 108 [101 to 114]
  Week 6 (V14) | 117 [113 to 122] | 124 [118 to 130] | 120 [113 to 128] | 122 [116 to 128] | 111 [94.0 to 129]
  Week 10 (V28) | 117 [111 to 122] | 121 [113 to 128] | 113 [107 to 119] | 124 [117 to 131] | 110 [101 to 119]
  Week 12 (V43): number analyzed (Participants) | 21 | 19 | 12 | 21 | 5
  Week 12 (V43) | 116 [112 to 121] | 119 [112 to 126] | 116 [108 to 124] | 122 [115 to 129] | 109 [101 to 117]

29. Primary Outcome: Resting Pulse Rate
Description: To measure resting heart rate in bpm.
Time Frame: Measured at Baseline (V3), week 6 (V14), week 10 (V28), and week 12 (V43).
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: beats/minute
Arm/Group | Cigarette Smoking | IQOS-1 | IQOS-2 | Smoking Abstinence | Other
Number analyzed (Participants) | 21 | 19 | 13 | 22 | 5
beats/minute
  Baseline (V3) | 68.8 [64.5 to 73.2] | 68.2 [63.8 to 72.5] | 67.9 [61.8 to 74.0] | 65.8 [61.0 to 70.5] | 73.8 [60.3 to 87.3]
  Week 6 (V14) | 65.1 [62.5 to 67.7] | 60.0 [56.5 to 63.5] | 63.3 [58.9 to 67.7] | 60.1 [56.3 to 63.9] | 62.2 [51.4 to 73.0]
  Week 10 (V28) | 65.1 [62.1 to 68.2] | 60.3 [56.4 to 64.3] | 60.7 [54.6 to 66.8] | 59.9 [56.0 to 63.8] | 65.4 [50.8 to 80.0]
  Week 12 (V43): number analyzed (Participants) | 21 | 19 | 12 | 21 | 5
  Week 12 (V43) | 70.5 [65.6 to 75.3] | 65.8 [61.4 to 70.2] | 69.5 [63.7 to 75.3] | 63.9 [59.2 to 68.6] | 73.2 [55.2 to 91.2]

30. Primary Outcome: Body Fat
Description: To measure body fat as a percentage.
Time Frame: Measured at Baseline (V3), at week 1 (V4), and at week 12 (V43).
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: % (body fat)
Arm/Group | Cigarette Smoking | IQOS-1 | IQOS-2 | Smoking Abstinence | Other
Number analyzed (Participants) | 21 | 19 | 13 | 22 | 5
% (body fat)
  Baseline (V3) | 27.8 [24.8 to 30.8] | 28.2 [24.6 to 31.8] | 25.6 [20.9 to 30.2] | 27.3 [23.2 to 31.5] | 20.5 [14.2 to 26.8]
  Acute Effect (V4) | 28.1 [25.3 to 30.9] | 28.6 [24.7 to 32.6] | 25.4 [19.6 to 31.2] | 28.1 [24.5 to 31.7] | 28 [20.7 to 35.3]
  Training Effect (V43): number analyzed (Participants) | 21 | 19 | 12 | 21 | 5
  Training Effect (V43) | 30.6 [27.5 to 33.7] | 27.5 [24.3 to 30.8] | 28 [23 to 33] | 29.9 [25.9 to 34] | 30.1 [23.1 to 37.2]

31. Primary Outcome: Waist Circumference
Description: To measure waist circumference in cm.
Time Frame: Measured at Baseline (V3), at week 1 (V4), and at week 12 (V43).
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: cm
Arm/Group | Cigarette Smoking | IQOS-1 | IQOS-2 | Smoking Abstinence | Other
Number analyzed (Participants) | 21 | 19 | 13 | 22 | 5
cm
  Baseline (V3) | 82.6 [77.9 to 87.3] | 83.7 [79 to 88.5] | 84.4 [80 to 88.8] | 84.9 [80.3 to 89.5] | 78.4 [63.5 to 93.3]
  Acute Effect (V4): number analyzed (Participants) | 17 | 14 | 12 | 19 | 5
  Acute Effect (V4) | 82.1 [76.6 to 87.5] | 81.6 [76.8 to 86.4] | 83.6 [77.7 to 89.5] | 85.2 [80.4 to 90.1] | 77.6 [63.5 to 91.7]
  Training Effect (V43): number analyzed (Participants) | 18 | 14 | 8 | 17 | 3
  Training Effect (V43) | 85.8 [80.5 to 91.1] | 86.6 [80.2 to 93.1] | 87.3 [78.3 to 96.2] | 89.5 [84.1 to 94.9] | 86 [54.9 to 117]

32. Primary Outcome: Body Weight
Description: To measure body weight in kilograms.
Time Frame: Measured at each visit, starting from Baseline (V3) until week 12 (V43).
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: kg
Arm/Group | Cigarette Smoking | IQOS-1 | IQOS-2 | Smoking Abstinence | Other
Number analyzed (Participants) | 21 | 19 | 13 | 22 | 5
kg
  Baseline (V3) | 72 [66.9 to 77.1] | 75.7 [69.7 to 81.7] | 75.5 [68.7 to 82.3] | 77.5 [72.2 to 82.8] | 69.3 [57.4 to 81.2]
  Acute Effect (V4) | 72.2 [67 to 77.4] | 75.7 [69.7 to 81.6] | 75.5 [68.5 to 82.4] | 77.6 [72.2 to 83] | 69.6 [57.5 to 81.7]
  Month 1 (V5 - V13) | 72 [66.9 to 77] | 75.7 [69.8 to 81.6] | 75.7 [69 to 82.5] | 77.9 [72.4 to 83.3] | 69.8 [57.3 to 82.2]
  Month 2 (V14 - V27) | 72 [67.1 to 76.8] | 75.8 [69.7 to 81.9] | 76.1 [69.4 to 82.9] | 78.1 [72.6 to 83.6] | 70.2 [57.2 to 83.1]
  Month 3 (V28 - V43) | 72 [67.1 to 76.8] | 75.8 [69.7 to 81.9] | 76.6 [69.6 to 83.5] | 78.3 [72.8 to 83.8] | 70.5 [57.8 to 83.2]

33. Primary Outcome: Exhaled Carbon Monoxide
Description: To measure exhaled carbon monoxide (ppm).
Time Frame: Measured at each visit, starting from Baseline (V3) until week 12 (V43).
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: ppm
Arm/Group | Cigarette Smoking | IQOS-1 | IQOS-2 | Smoking Abstinence | Other
Number analyzed (Participants) | 21 | 19 | 13 | 22 | 5
ppm
  Baseline (V3) | 20.8 [17.3 to 24.3] | 20.8 [16.6 to 25.0] | 19.7 [14.8 to 24.6] | 18.6 [14.7 to 22.6] | 20.4 [7.30 to 33.5]
  Week 1 (V4) | 25.4 [20.7 to 30.1] | 6.16 [2.44 to 9.87] | 5.46 [2.36 to 8.56] | 3.55 [2.53 to 4.56] | 4.80 [-0.274 to 9.87]
  Week 6 (V14) | 20.6 [15.3 to 25.9] | 5.00 [2.84 to 7.16] | 8.38 [-3.78 to 20.6] | 2.77 [2.32 to 3.23] | 2.60 [0.717 to 4.48]
  Week 10 (V28) | 20.6 [16.3 to 24.9] | 4.58 [2.69 to 6.47] | 4.00 [2.60 to 5.40] | 2.64 [2.05 to 3.23] | 2.40 [0.984 to 3.82]
  Week 12 (V43): number analyzed (Participants) | 21 | 19 | 12 | 21 | 5
  Week 12 (V43) | 21.8 [16.8 to 26.7] | 5.79 [2.96 to 8.62] | 3.17 [1.52 to 4.81] | 3.05 [2.14 to 3.95] | 2.00 [0.758 to 3.24]

34. Primary Outcome: Carboxyhemoglobin
Description: To measure Carboxyhemoglobin (COHb), assayed from whole blood. Expressed as % of saturation of hemoglobin.
Time Frame: Measured at Baseline (V3), week 1 (V4), week 6 (V14), week 10 (V28), and week 12 (V43).
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: % (of saturation of hemoglobin)
Arm/Group | Cigarette Smoking | IQOS-1 | IQOS-2 | Smoking Abstinence | Other
Number analyzed (Participants) | 21 | 19 | 13 | 22 | 5
% (of saturation of hemoglobin)
  Baseline (V3): number analyzed (Participants) | 21 | 19 | 13 | 22 | 4
  Baseline (V3) | 1.92 [1.43 to 2.58] | 2.37 [1.82 to 3.09] | 1.71 [1.31 to 2.23] | 1.74 [1.10 to 2.74] | 2.50 [1.10 to 5.69]
  Week 1 (V4) | 3.29 [2.61 to 4.16] | 0.422 [0.231 to 0.773] | 0.372 [0.151 to 0.915] | 0.272 [0.163 to 0.456] | 0.426 [0.172 to 1.06]
  Week 6 (V14) | 2.51 [1.99 to 3.16] | 0.350 [0.181 to 0.679] | 0.109 [0.0509 to 0.234] | 0.110 [0.0703 to 0.173] | 0.272 [0.0778 to 0.954]
  Week 10 (V28) | 3.01 [2.34 to 3.87] | 0.338 [0.190 to 0.601] | 0.285 [0.158 to 0.513] | 0.189 [0.128 to 0.279] | 0.432 [0.0520 to 3.58]
  Week 12 (V43): number analyzed (Participants) | 21 | 19 | 12 | 21 | 5
  Week 12 (V43) | 2.04 [1.60 to 2.61] | 0.187 [0.0868 to 0.402] | 0.0674 [0.0395 to 0.115] | 0.0864 [0.0557 to 0.134] | 0.132 [0.0495 to 0.352]

35. Primary Outcome: NEQ
Description: To measure Nicotine equivalents (NEQ) concentrations, measured in spot urine and expressed as concentration adjusted for creatinine.
Time Frame: Measured at Baseline (V3), week 1 (V4), week 6 (V14), week 10 (V28), and week 12 (V43).
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: mg/g creat
Arm/Group | Cigarette Smoking | IQOS-1 | IQOS-2 | Smoking Abstinence | Other
Number analyzed (Participants) | 21 | 19 | 13 | 22 | 5
mg/g creat
  Baseline (V3) | 14.9 [11.7 to 19.0] | 14.2 [11.5 to 17.5] | 10.5 [7.55 to 14.5] | 12.9 [10.1 to 16.3] | 14.0 [6.14 to 32.1]
  Week 1 (V4) | 13.2 [10.2 to 17.0] | 10.9 [7.90 to 15.0] | 7.08 [4.38 to 11.5] | 4.40 [2.36 to 8.18] | 8.49 [1.39 to 51.9]
  Week 6 (V14) | 13.2 [10.2 to 17.0] | 10.9 [7.90 to 15.0] | 7.08 [4.38 to 11.5] | 4.40 [2.36 to 8.18] | 9.03 [1.19 to 68.6]
  Week 10 (V28): number analyzed (Participants) | 21 | 19 | 13 | 21 | 5
  Week 10 (V28) | 14.3 [12.2 to 16.6] | 11.4 [7.94 to 16.4] | 8.66 [5.27 to 14.2] | 1.59 [0.774 to 3.25] | 11.6 [1.93 to 70.2]
  Week 12 (V43): number analyzed (Participants) | 21 | 19 | 12 | 21 | 5
  Week 12 (V43) | 13.8 [11.4 to 16.8] | 12.3 [9.69 to 15.7] | 5.93 [3.86 to 9.11] | 2.70 [1.49 to 4.90] | 5.87 [1.28 to 27.0]

36. Primary Outcome: Total NNAL
Description: To measure Total 4-(methylnitrosamino)-1-(3-pyridyl)-1-butanol (NNAL) concentrations, measured in spot urine and expressed as concentration adjusted for creatinine.
Time Frame: Measured at Baseline (V3), week 1 (V4), week 6 (V14), week 10 (V28), and week 12 (V43).
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: pg/mg creat
Arm/Group | Cigarette Smoking | IQOS-1 | IQOS-2 | Smoking Abstinence | Other
Number analyzed (Participants) | 21 | 19 | 13 | 22 | 5
pg/mg creat
  Baseline (V3) | 170 [99.3 to 291] | 239 [184 to 310] | 164 [87.5 to 307] | 166 [114 to 243] | 244 [73.3 to 813]
  Week 1 (V4) | 147 [84.5 to 254] | 88.3 [45.8 to 170] | 69.9 [31.9 to 153] | 45.8 [30.6 to 68.5] | 97.9 [38.0 to 252]
  Week 6 (V14) | 177 [113 to 278] | 90.2 [62.6 to 130] | 62.7 [31.8 to 123] | 17.4 [9.53 to 31.9] | 93.4 [30.7 to 284]
  Week 10 (V28) | 221 [155 to 315] | 81.3 [49.3 to 134] | 74.6 [32.4 to 171] | 26.1 [12.1 to 56.4] | 83.3 [14.1 to 490]
  Week 12 (V43): number analyzed (Participants) | 21 | 19 | 12 | 21 | 5
  Week 12 (V43) | 214 [163 to 280] | 82.5 [46.1 to 148] | 37.9 [20.7 to 69.4] | 41.3 [22.9 to 74.5] | 62.3 [21.3 to 182]

37. Primary Outcome: CEMA
Description: To measure 2-cyanoethylmercapturic acid (CEMA) concentrations, measured in spot urine and expressed as concentration adjusted for creatinine.
Time Frame: Measured at Baseline (V3), week 1 (V4), week 6 (V14), week 10 (V28), and week 12 (V43).
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mg creat
Arm/Group | Cigarette Smoking | IQOS-1 | IQOS-2 | Smoking Abstinence | Other
Number analyzed (Participants) | 21 | 19 | 13 | 22 | 5
ng/mg creat
  Baseline (V3) | 140 [106 to 185] | 170 [143 to 202] | 135 [97.1 to 188] | 128 [95.9 to 172] | 144 [57.3 to 362]
  Week 1 (V4) | 147 [114 to 189] | 39.5 [26.8 to 58.4] | 28.1 [14.6 to 53.9] | 25.3 [18.3 to 34.9] | 37.5 [12.9 to 109]
  Week 6 (V14) | 139 [104 to 185] | 26.6 [15.8 to 44.8] | 15.3 [7.89 to 29.8] | 12.1 [8.47 to 17.2] | 33.1 [6.10 to 180]
  Week 10 (V28) | 148 [113 to 194] | 23.6 [14.4 to 38.7] | 12.7 [5.99 to 26.9] | 11.0 [7.58 to 15.9] | 19.3 [4.88 to 76.0]
  Week 12 (V43): number analyzed (Participants) | 21 | 19 | 12 | 21 | 5
  Week 12 (V43) | 141 [108 to 183] | 24.8 [12.4 to 49.4] | 8.67 [4.05 to 18.6] | 12.7 [7.50 to 21.3] | 16.5 [3.90 to 69.7]

38. Primary Outcome: Nicotine/Tobacco Product Use (Cigarettes)
Description: To measure self-reported number of any nicotine/tobacco product used on a daily basis.
Time Frame: Recorded daily by subject, in product use diary, from study enrollment for 16 weeks.
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: cigarettes per day
Arm/Group | Cigarette Smoking | IQOS-1 | IQOS-2 | Smoking Abstinence | Other
Number analyzed (Participants) | 21 | 19 | 13 | 22 | 5
cigarettes per day
  Pre-randomization (V2-V3): number analyzed (Participants) | 17 | 18 | 12 | 22 | 3
  Pre-randomization (V2-V3) | 16.8 [13.9 to 19.7] | 19.0 [16.4 to 21.5] | 17.4 [14.3 to 20.4] | 17.7 [14.7 to 20.8] | 24.1 [18.9 to 29.4]
  Week 1 (V3-V4): number analyzed (Participants) | 19 | 19 | 13 | 21 | 3
  Week 1 (V3-V4) | 17.5 [15.0 to 20.0] | 0.206 [0 to 0.439] | 0.242 [0 to 0.556] | 0.0136 [0 to 0.0420] | 9.72 [0 to 41.4]
  Up to month 1 (V3-V14): number analyzed (Participants) | 21 | 19 | 13 | 22 | 4
  Up to month 1 (V3-V14) | 17.3 [15.2 to 19.5] | 0.0351 [0 to 0.0753] | 0.0623 [0 to 0.132] | 0.00222 [0 to 0.00683] | 8.86 [0 to 25.0]
  Up to month 2 (V3-V26: number analyzed (Participants) | 21 | 19 | 13 | 22 | 4
  Up to month 2 (V3-V26 | 17.1 [14.8 to 19.4] | 0.0196 [0 to 0.0413] | 0.0369 [0 to 0.0783] | 0.00132 [0 to 0.00406] | 8.38 [0 to 24.3]
  Overall (V3-V43): number analyzed (Participants) | 21 | 19 | 13 | 22 | 4
  Overall (V3-V43) | 17.1 [14.7 to 19.5] | 0.0142 [0.000387 to 0.0280] | 0.0273 [0 to 0.0592] | 0.000858 [0 to 0.00264] | 8.34 [0 to 24.3]

39. Primary Outcome: Nicotine/Tobacco Product Use (HeatSticks)
Description: To measure self-reported number of any nicotine/tobacco product used on a daily basis.
Time Frame: Recorded daily by subject, in product use diary, from study enrollment for 16 weeks.
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: heatsticks per day
Arm/Group | Cigarette Smoking | IQOS-1 | IQOS-2 | Smoking Abstinence | Other
Number analyzed (Participants) | 21 | 19 | 13 | 22 | 5
heatsticks per day
  Pre-randomization (V2-V3): number analyzed (Participants) | 17 | 18 | 12 | 22 | 3
  Pre-randomization (V2-V3) | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
  Week 1 (V3-V4): number analyzed (Participants) | 19 | 19 | 13 | 21 | 3
  Week 1 (V3-V4) | 0 [0 to 0] | 17.7 [13.3 to 22.1] | 14.1 [10.5 to 17.7] | 0 [0 to 0] | 5.81 [0 to 30.8]
  Up to month 1 (V3-V14): number analyzed (Participants) | 21 | 19 | 13 | 22 | 4
  Up to month 1 (V3-V14) | 0 [0 to 0] | 18.6 [14.4 to 22.9] | 14.0 [10.8 to 17.1] | 0 [0 to 0] | 4.97 [0 to 20.8]
  Up to month 2 (V3-V26: number analyzed (Participants) | 21 | 19 | 13 | 22 | 4
  Up to month 2 (V3-V26 | 0 [0 to 0] | 18.7 [14.5 to 22.9] | 14.1 [10.9 to 17.4] | 0 [0 to 0] | 4.97 [0 to 20.8]
  Overall (V3-V43): number analyzed (Participants) | 21 | 19 | 13 | 22 | 4
  Overall (V3-V43) | 0 [0 to 0] | 19.0 [14.6 to 23.3] | 14.1 [10.9 to 17.2] | 0 [0 to 0] | 5.08 [0 to 21.3]

40. Primary Outcome: Nicotine/Tobacco Product Use (E-cigarettes)
Description: To measure self-reported number of any nicotine/tobacco product used on a daily basis.
Time Frame: Recorded daily by subject, in product use diary, from study enrollment for 16 weeks.
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: e-cigarettes per day
Arm/Group | Cigarette Smoking | IQOS-1 | IQOS-2 | Smoking Abstinence | Other
Number analyzed (Participants) | 21 | 19 | 13 | 22 | 5
e-cigarettes per day
  Pre-randomization (V2-V3): number analyzed (Participants) | 17 | 18 | 12 | 22 | 3
  Pre-randomization (V2-V3) | 0 [0 to 0] | 0 [0 to 0] | 0.0952 [0 to 0.305] | 0 [0 to 0] | 0 [0 to 0]
  Week 1 (V3-V4): number analyzed (Participants) | 19 | 19 | 13 | 21 | 3
  Week 1 (V3-V4) | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
  Up to month 1 (V3-V14): number analyzed (Participants) | 21 | 19 | 13 | 22 | 4
  Up to month 1 (V3-V14) | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
  Up to month 2 (V3-V26: number analyzed (Participants) | 21 | 19 | 13 | 22 | 4
  Up to month 2 (V3-V26 | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
  Overall (V3-V43): number analyzed (Participants) | 21 | 19 | 13 | 22 | 4
  Overall (V3-V43) | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the signature of the ICF by each subject until the end of the safety follow-up period, for a total study duration of up to 24 weeks for each subject.
Description: The safety set comprised the 93 subjects enrolled in the study. Adverse events are reported according to the study arm (Cigarette; IQOS-1; IQOS-2; and Smoking Abstinence) that each subject was randomized to.
Groups:
- Other: Other product use (use of <30 HeatSticks/month and 5-30 cig/month or other forms of product use)
Arm/Group | Cigarette Smoking | IQOS-1 | IQOS-2 | Smoking Abstinence | Other
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/22 | 0/13 | 0/24 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22 | 1/13 | 1/24 | 0/12
Other Adverse Events (participants affected / at risk) | 12/22 | 10/22 | 8/13 | 12/24 | 5/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cigarette Smoking (N=22) | IQOS-1 (N=22) | IQOS-2 (N=13) | Smoking Abstinence (N=24) | Other (N=12)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cigarette Smoking (N=22) | IQOS-1 (N=22) | IQOS-2 (N=13) | Smoking Abstinence (N=24) | Other (N=12)
Nasopharyngitis (Infections and infestations) | 8 (8) | 3 (3) | 3 (3) | 3 (3) | 3 (3)
Gastroenteritis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Blood Tryglycerides Increased (Investigations) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 1 (2) | 0 (0) | 1 (1) | 4 (4) | 1 (1)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
We confirm we have the contractual provisions in place which specify that in no event will the study site be allowed to disclose to any third party (or publicly release) any information obtained through the study without the CRO's prior written consent which in turn cannot provide such consent without Sponsor's approval unless such publication is made to satisfy regulatory requirements.

The Intellectual Property rights and research results from the present study belong to the Sponsor.

DOCUMENTS (2):
  • Study Protocol (2019-05-02): https://cdn.clinicaltrials.gov/large-docs/17/NCT03887117/Prot_000.pdf
  • Statistical Analysis Plan (2020-03-10): https://cdn.clinicaltrials.gov/large-docs/17/NCT03887117/SAP_001.pdf